CLINICAL TRIAL: NCT05538845
Title: Comparison of Screw and Suture Button Technique Results in Ankle Syndesmosis Injuries
Status: Completed | Type: Observational
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Yusuf Sait Durak, Principal Investigator,, Ataturk University
Other Study IDs: atauni orthopedia ankle
Record Dates: First submitted 2022-08-25; First posted 2022-09-14 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Ankle Injuries; Syndesmotic Injuries; Tibiofibular; Dislocation Distal
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Screw: Screw fixation
  Interventions: Device: Screw fixation
- Suture button: Suture button
  Interventions: Device: Suture button

INTERVENTIONS:
Device: Screw fixation — Screw fixation to patients
  Groups: Screw
Device: Suture button — Suture button for patients
  Groups: Suture button

SUMMARY:
In this study, syndesmosis injuries were detected in 143 of the patients who came to Atatürk University Faculty of Medicine, Orthopedics and Traumatology clinic from October 2017 to October 2021 with ankle fractures. 33 of these patients couldn't followed for various reasons. Screw or suture buttone method was applied on 110 patients. And patients were examined with lots of data to compare their results. A retrospective study was conducted.

ELIGIBILITY:
Inclusion Criteria:

* Ankle fractures associated with syndesmotic injury
* Age group 19-91 years
* Dislocation or non-dislocation ankle fractures
* Fractures due to acute injury (less than 3 weeks)
* Patient compliance with follow-up

Exclusion Criteria:

* Patients younger than 18 years of age
* Conservative treatment
* Pathological and neglected fractures
* Patient's non-compliance with follow-up

Ages: 19 Years to 91 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Comparison of 110 patients with screw or suture button method.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
angles of the joint range of motion | 12 months after surgery
  Calculate joint range of motion by measuring the angles between the beginning position and the ending position of available motion with goniometer

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University School of Medicine, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hennings R, Fuchs C, Spiegl UJ, Theopold J, Souleiman F, Kleber C, Ahrberg AB. "Flexible nature of fixation" in syndesmotic stabilization of the inferior tibiofibular joint affects the radiological reduction outcome. Int Orthop. 2022 Nov;46(11):2649-2657. doi: 10.1007/s00264-022-05550-7. Epub 2022 Aug 19. PMID 35982324
- [Background] Hakverdiyev Y, McFarland EG, Kaymakoglu M, Ozdemir E, Akpinar S, Huri P, Costouros JG, Huri G. Biomechanical Strength of Screw Versus Suture Button Fixation in the Latarjet Procedure: A Cadaver Study. Orthopedics. 2022 Nov-Dec;45(6):e321-e325. doi: 10.3928/01477447-20220805-01. Epub 2022 Aug 10. PMID 35947455